CLINICAL TRIAL: NCT03072719
Title: A Clinical Study Investigating the Efficacy of a Dentifrice in Providing Immediate and Short Term Relief From Dentinal Hypersensitivity
Brief Title: The Efficacy of a Dentifrice in Providing Relief From Immediate and Short Term Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202161; RH01327 (Other: GSK); NCT01724008 (obsolete NCT alias)
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2017-04-18 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dentifrice containing stannous fluoride (Experimental): Toothpaste
  Interventions: Drug: Stannous Fluoride
- Dentifrice containing Sodium Monofluorophosphate (Active Comparator): Toothpaste
  Interventions: Drug: Sodium Monofluorophosphate

INTERVENTIONS:
Drug: Stannous Fluoride — Test dentifrice, participants will brush each of the 2 selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least one minute.
  Arms: Dentifrice containing stannous fluoride
Drug: Sodium Monofluorophosphate — Control dentifrice, participants will brush the whole mouth thoroughly for at least 1 minute.
  Arms: Dentifrice containing Sodium Monofluorophosphate

SUMMARY:
A randomised, examiner blind, two treatment arm, stratified, parallel design, single-site study in subjects with at least two sensitive teeth to compare the efficacy of a test dentifrice against that of a control dentifrice in reducing dentinal hypersensitivity.

ELIGIBILITY:
Inclusion

* Demonstrates understanding of the study and willingness to participate
* Aged at least 18 to 65 years
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral examination.
* Self-reported history of dentinal hypersensitivity lasting more than 6 months but not more than 10 years
* Minimum of 20 natural teeth at screening, a minimum of two accessible teeth (incisors, canines, pre-molars)
* At baseline, participant has two non-adjacent sensitive teeth from those meeting the EAR, GI and mobility criteria at screening, with sensitivity measured by tactile stimulus (Yeaple ≤ 20g) and evaporative (air) assessment (Schiff Sensitivity Score ≥ 2) at baseline

Exclusion

* Pregnant or breast-feeding women
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia
* Dental prophylaxis within 4 weeks of screening
* Tongue or lip piercing or presence of dental implants
* Professional desensitising treatment within 12 weeks of screening
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening.
* Teeth bleaching within 12 weeks of screening
* Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine
* Sensitive tooth not expected to respond to treatment with an over-the counter dentifrice in the opinion of the investigator.
* Use of a desensitising dentifrice within six weeks of screening (participant will be required to bring their current dentifrice to the site in order to verify the lack of known anti-sensitivity ingredients)
* Daily doses of a medication which, in the opinion of the investigator, could interfere with the perception of pain
* Currently taking antibiotics or have taken antibiotics within 2 weeks of baseline.
* Daily doses of a medication which, in the opinion of the investigator, causes xerostomia
* Individuals who require antibiotic prophylaxis for dental procedures
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cork, Ireland

REFERENCES:
- [Derived] Parkinson CR, Hughes N, Hall C, Whelton H, Gallob J, Mason S. Three randomized clinical trials to assess the short-term efficacy of anhydrous 0.454% w/w stannous fluoride dentifrices for the relief of dentin hypersensitivity. Am J Dent. 2016 Feb;29(1):25-32. PMID 27093773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in Ireland.
Pre-assignment Details: Total 394 participants were screened, out of which 120 participants were randomized. 274 participants were not randomized because 248 participants did not meet the study criteria, 4 participants were lost to follow up, and 7 participants withdrew the consent and 15 participants for other reasons (not-specified).
Groups:
- Experimental Dentifrice: Participants were instructed to dose a dry toothbrush with at least a 1-inch strip of the experimental dentifrice (0.454% Stannous Fluoride, 1100 parts per million [ppm] as fluoride) and then to brush each of the 2 selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least 1 minute.
- Reference Dentifrice: Participants were instructed to dose a dry toothbrush according to their normal habit with reference dentifrice (0.76% sodium monofluorophosphate, 1000ppm as fluoride) and brushed the whole mouth thoroughly (as per the manufacturer's instructions), for at least 1 minute.
Period: Overall Study
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Started | 60 | 60
Completed | 59 | 59
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental Dentifrice: Participants were instructed to dose a dry toothbrush with at least a 1-inch strip of the experimental dentifrice (0.454% Stannous Fluoride, 1100ppm as fluoride) and then to brush each of the 2 selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least 1 minute.
- Total: Total of all reporting groups
Arm/Group | Experimental Dentifrice | Reference Dentifrice | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.4 (12.85) | 30.7 (11.66) | 29.5 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 75
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 59 | 59 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 60 | 59 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 14
Description: Schiff sensitivity score was assessed by examiner as participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth. Response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity.
Time Frame: Baseline, Day 14
Population: Analysis for this outcome was conducted on intent-to-treat (ITT) population which included all randomized participants who had at least one post baseline assessment of efficacy. n is the number of participants evaluated at specific time point for treatment arms respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 60 | 60
score on a scale
  At Baseline | 2.51 (0.437) | 2.51 (0.446)
  At Day 14: number analyzed (Participants) | 59 | 59
  At Day 14 | 1.16 (0.774) | 1.35 (0.901)
  Change from Baseline on Day 14: number analyzed (Participants) | 59 | 59
  Change from Baseline on Day 14 | -1.35 (0.727) | -1.16 (0.762)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; H0 : The difference in Schiff Sensitivity Score at Day 14 between the experimental dentifrice and reference dentifrice is zero. H1 : The difference in Schiff Sensitivity Score at Day 14 between the experimental dentifrice and reference dentifrice is not zero; Test type: Superiority or Other; p = 0.1774, ANCOVA — From ANCOVA model: Treatment as fixed factor, baseline Schiff Sensitivity score as covariate; Least square (LS) mean difference = -0.19, 95% CI 2-sided [-0.46 to 0.09] — Difference is 0.454% stannous fluoride minus 0.76% sodium monofluorophosphate such that a negative difference favours first named treatment

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score on Post First Brushing (After 5 Minutes) and Day 3
Description: Schiff sensitivity score was assessed by examiner as participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth. Response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity.
Time Frame: Baseline, post first brushing (after 5 minutes) and Day 3
Population: Analysis for this outcome was conducted on ITT population which included all randomized participants who had at least one post baseline assessment of efficacy. n is the number of participants evaluated at specific time points for treatment arms respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 60 | 60
score on a scale
  After 5 minutes of brushing | 1.73 (0.826) | 1.92 (0.737)
  Change after 5 minutes of brushing | -0.78 (0.660) | -0.59 (0.571)
  On Day 3: number analyzed (Participants) | 54 | 57
  On Day 3 | 1.63 (0.784) | 1.77 (0.785)
  Change from baseline on Day 3: number analyzed (Participants) | 54 | 57
  Change from baseline on Day 3 | -0.88 (0.658) | -0.74 (0.568)

3. Secondary Outcome: Change From Baseline in Tactile (Yeaple) Pain Threshold on Post First Brushing (After 5 Minutes), Day 3 and Day 14
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline, post first brushing (after 5 minutes), Day 3 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 60 | 60
gram (g)
  At Baseline | 10.8 (2.29) | 11.5 (2.65)
  After 5 minutes of brushing | 16.5 (13.82) | 16.7 (11.19)
  Change after 5 minutes of brushing | 5.7 (13.45) | 5.2 (10.93)
  On Day 3: number analyzed (Participants) | 57 | 60
  On Day 3 | 18.4 (17.32) | 18.6 (16.73)
  Change from baseline on Day 3: number analyzed (Participants) | 57 | 60
  Change from baseline on Day 3 | 7.5 (17.73) | 7.1 (16.48)
  On Day 14: number analyzed (Participants) | 59 | 59
  On Day 14 | 25.3 (22.64) | 23.8 (22.33)
  Change from baseline on Day 14: number analyzed (Participants) | 59 | 59
  Change from baseline on Day 14 | 14.6 (22.67) | 12.3 (21.68)

ADVERSE EVENTS:
Arm/Group | Experimental Dentifrice | Reference Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 9/60 | 8/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Dentifrice (N=60) | Reference Dentifrice (N=60)
Sensitivity of Teeth (Gastrointestinal disorders) | 5 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Tooth Injury (Injury, poisoning and procedural complications) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Axillary Candidiasis (Infections and infestations) | 1 | 0
Axillary Pain (General disorders) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.